CLINICAL TRIAL: NCT05288049
Title: Treating Early Stages Of seveRe Mental disOrders With an Intervention Targeting Cognitive Reserve
Brief Title: Treating Early Stages With an Intervention Targeting Cognitive Reserve
Acronym: TESORO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCLinic
Record Dates: First submitted 2021-12-08; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2021-12

CONDITIONS: Psychotic Disorder
Keywords: cognitive reserve; psychotic disorder; offsprings
MeSH Terms: conditions — Psychotic Disorders | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: An experimental randomized controlled clinical study is proposed, which will be rater-blinded and stratified by age, gender and socioeconomic status to assess the efficacy of a new intervention designed to increase CR in FEP and HR-SZBD subjects.
Who Masked: Investigator
Masking Description: The experimental group will receive 12 weekly sessions (1 per week) of the intervention, which will be conducted by two psychologists blinded to the assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention aiming to enhance cognitive reserve (CR) (Experimental): The psychological intervention to enhance cognitive reserve (CR) will be conducted in a group format (6-8 individuals). Each session will last approximately 60 minutes. The full psychological intervention will have 12 sessions (1 per week) and will last three months. Moreover, to remind the participants of the contents of the intervention, a follow-up session will be held every two months between the last session of the psychological intervention and the 12-month assessment. Most of the tasks of the psychological intervention will use pen and paper with audiovisual support. However, some sessions will use mobile apps and virtual reality. Virtual reality will be implemented for each patient in the sessions focusing on mindfulness training. The contents of the sessions are adapted to the different ages of the attendees. Groups with adolescents and those with young adults will be run separately.
  Interventions: Behavioral: Enhancing cognitive reserve
- Support therapy (Active Comparator): The support control group will have weekly meetings with assistants to talk about the difficulties they had during the week, without receiving a specific intervention. After the 12-month assessment, subjects in the support group will be offered the intervention although this will be out of the scope of this study.
  Interventions: Behavioral: Support therapy

INTERVENTIONS:
Behavioral: Enhancing cognitive reserve — The CR enhancement protocol consists of 12 weekly sessions in a group format with audiovisual and technological devices support. All sessions are held separately for parents and children, adolescents and young adults. All material is adapted to different ranges of age. This same protocol will be adapted for patients with a first affective or non-affective episode. Two sessions are about to promote healthy lifestyle by implementing healthy habits, two more sessions about training and practice mindfulness with virtual reality devices, two sessions about improving leisure-time activities, focused on promoting of intellectual and/or cultural activities as leisure time as well as physical exercise, the rest of sessions are about to promote vocational and educational activities, metacognition, social skills, problem-solving techniques and how to detect and act on warning signs, a brief psychoeducative session about the main early warning signs of general psychopathology.
  Arms: Intervention aiming to enhance cognitive reserve (CR)
Behavioral: Support therapy — The support control group will have weekly meetings with assistants to talk about the difficulties they had during the week, without receiving a specific intervention.
  Arms: Support therapy

SUMMARY:
This study proposes continuity in the implementation of a psychological approach program to enhance cognitive reserve (CR) in children, adolescent and young adults, off-springs of patients with schizophrenia or bipolar disorder (Off-SZBP), and first affective and non-affective episodes with three main objectives: to characterize the cognitive reserve in the early stages of the disease, to validate the adaptation of the intervention to first affective and non-affective disorders to assess the effectiveness of the intervention in a longer term.

DETAILED DESCRIPTION:
The study will include a sample of High Genetic Risk-SZBD (HR-SZBD) subjects (N = 60), First Episode Psychotic Patients (FEP) (N = 60) and CC participants (N = 60). All groups will be evaluated with CR scales as well as clinical, neuropsychological, and neuroimaging tests at baseline. The FEP and HR-SZBD groups will then be randomly allocated to a psychological intervention to enhance CR (N = 30 FEP and 30 HR-SZBD) or a support group (N = 30 FEP and 30 HR-SZBD). Once the psychological intervention (3 months) is completed, the FEP and HR-SZBD groups will be re-assessed with the same clinical, neuropsychological, and neuroimaging tests as well as CR scales that were used at baseline. Between the third and twelfth month, follow-up sessions will be conducted to remind the participants of the contents of the intervention. Finally, clinical, CR, neuropsychological and neuroimaging assessments will be completed in the FEP, HR-SZBD and CC groups at 12 months to verify whether the effects of the intervention remain stable over time.

ELIGIBILITY:
Inclusion Criteria:

1. - Inclusion criteria for the Off-SZBP will be: Subjects between 12 and 25 years with a parent (mother or father) diagnosed with bipolar disorder or schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria.
2. - Inclusion criteria for patients with a first affective (mania or depression with or without psychotic symptoms and hypomania) or non-affective episode (first psychotic episode) will be:

   1. Patients between 12 and 45 years with a first affective or non-affective episode within the last 5 years.
   2. Diagnosis of bipolar disorder, schizophrenia, schizoaffective disorders and other psychoses according to DSM-5 criteria based on a semi-structured clinical interview.
   3. Patients in full or partial clinical remission at the moment of assessment, defined as scores ≤ 10 in Young Mania Rating Scale (YMRS) (Young, 1978) and ≤ 14 scores in the Hamilton Depression Rating Scale (Hamilton, 1960).
   4. Scores lower or equal to 3 during the previous two months in symptoms P1 (delusions), G9 (unusual thought content), P3 (hallucinations), P2 (conceptual disorganization), G5 (mannerisms and posturing), N1 (blunted affect), N4 (social withdrawal) and N6 (spontaneity and flow of conversation) on the scale for positive and negative schizophrenia syndrome (PANSS).
3. - Inclusion criteria for Community Control:s (CC) Children, adolescents and young adults between 12 and 45 years old without history of psychotic disorder or bipolar disorder in first degree relatives.

   * Exclusion criteria, common to all participants, will be:

     1. Estimated Intelligence quotient < 70.
     2. Any medical condition that could affect neuropsychological performance (such as neurological diseases) or history of head trauma with loss of consciousness.
     3. To have participated in any structured psychosocial intervention within the past 6 months.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
cognitive reserve | 12 months
  the enhancing of cognitive reserve by means of the Cognitive Reserve Assessment Scale (CRASH scale). The CRASh scale is an interviewer-administered instrument which consists of 23 items to assess three domains related with the cognitive reserve: education, occupation and leisure and intellectual activities. This last domain will have evaluated taking into account the different life stages (childhood/adolescence, adulthood and current situation). The scale provides a total score and different scores for each specific domain. The maximum total score is 60 points. Each domain scores is calculated by adding all items of the domain. The higher scores, the higher CR level.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No